CLINICAL TRIAL: NCT03097705
Title: The Effect of Steep Trendelenburg Position Used During Laparoscopic Surgery on Intraocular Pressure During Surgery and on the Retinal Nerve Fiber Thickness After Surgery
Brief Title: Effect of Steep Trendelenburg in Laparoscopic Surgery on IOP & RNFL Thickness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Orna Geyer, PROFESSOR, Carmel Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CMC-17-0026-CTIL
Record Dates: First submitted 2017-03-08; First posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Intraocular Pressure; Retinal Nerve Fiber Bundle Deficiency
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IOP and OCT RNFL measurements (Other): all subjects will undergo ophthalmological exams including IOP and RNFL OCT measurements
  Interventions: Diagnostic Test: OCT (Optical coherence tomography)

INTERVENTIONS:
Diagnostic Test: OCT (Optical coherence tomography) — RNFL AND IOP MEASUREMNTS
  Other Names: CARE (ICARE FINLAND Oy)

SUMMARY:
The effect of Steep Trendelenburg position used during laparoscopic surgery on intraocular pressure during surgery and on the retinal nerve fiber thickness after surgery

DETAILED DESCRIPTION:
To measure IOP and RNFL thickness in subjects undergoing laparoscopic operations in steep trendelenburg before, during, and after the operation

ELIGIBILITY:
Inclusion Criteria:

* SUBJECTS INTENDING TO UNDERGO LAPROSCOPIC SERGURY WHICH HAVE NO EYE DISEASES

Exclusion Criteria:

* SUBJECT WITH EYES DISEASE
* PREGNANCY DURING THE STUDY PERIOD

Ages: 40 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-04-20 (Estimated); Primary Completion 2017-09-12 (Estimated); Study Completion 2018-03-12 (Estimated)

PRIMARY OUTCOMES:
Intra Ocular Pressure (IOP) | Change in IOP from baseline to IOP during surgery and to one week and to three months following surgery
  IOP measurement will be taken before, during and after surgery using ICARE tonometer
Retinal Nerve Fiber Layer Thickness (RNFL) using OCT | Change in OCT RNFL thickness from baseline to OCT RNFL thickness during surgery and to one week and to three months following surgery
  RNFL measurement will be taken before and after surgery using spectralis OCT

IPD SHARING:
Plan to Share IPD: No